CLINICAL TRIAL: NCT01707212
Title: A Prenatal Education Module for Parents to Improve the Use of Pain-management Strategies for Immunization in Two-month Old Infants: a Randomized Controlled Trial of Knowledge Translation
Brief Title: Prenatal Education About Infant Immunization Pain Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, Anna Taddio, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0134-E
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Immunization
Keywords: parent education; pain management; immunization; infant
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain management education (Experimental): Education about pain management during infant immunization
  Interventions: Behavioral: Pain management education
- No pain management education (Other): Control - general information about immunization only
  Interventions: Behavioral: No pain management education

INTERVENTIONS:
Behavioral: Pain management education — Education about pain management during infant immunization
  Arms: Pain management education
Behavioral: No pain management education — Control - no education about pain management during infant immunization
  Arms: No pain management education

SUMMARY:
There are numerous pain management strategies available for the management of infant immunization pain. The majority of infants, however do not benefit from these interventions, which causes them to suffer pain unnecessarily. This study will assess the impact of educating parents about pain management strategies on their knowledge and behaviour regarding pain management during routine 2-month infant immunization injections.

DETAILED DESCRIPTION:
There is ample literature outlining effective pain management strategies for immunization including psychological, physical and pharmacological interventions; however their use in clinical practice has been limited. Teaching parents about these strategies in an enriching setting such as prenatal education classes has the potential to increase utilization of these strategies, and empower parents to take on a more active role in the management of their infant's pain during routine immunization. Educating parents about pain-management for infant immunization has not been previously investigated in this setting. The aim of this cluster-randomized controlled trial is to evaluate the effectiveness of an immunization pain-management education module added to the prenatal education program at Mount Sinai Hospital on parental knowledge and behaviour regarding pain management during routine 2-month infant immunization injections.

ELIGIBILITY:
Inclusion Criteria:

* mothers attending weekend prenatal classes
* delivery of a healthy newborn > 35 weeks gestational age
* available for followup for infant's 2-month immunization

Exclusion Criteria:

* mothers who do not plan to immunize their infants
* infant with major birth defect or hospitalized at time of immunization
* mothers who need to attend the prenatal class at a separate time when education not offered

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Utilization of pain management strategies during infant immunization | within 2 months of immunization
  Parents will self-report utilization of specific pain management strategies during routine 2-month infant immunization

SECONDARY OUTCOMES:
Attempted use of pain management strategies during infant immunization | within 2 months of immunization
  Parents will self-reported attempted utilization of specific pain management strategies at 2-month infant immunization
Knowledge | within 2 months of immunization
  Parents will answer questions regarding their knowledge about the effectiveness of various pain management strategies for infant immunization injections

OTHER OUTCOMES:
Infant pain during immunization | within 2 months of immunization
  Parents will self-report infant pain during 2-month immunization using an 11-point Numerical Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada